CLINICAL TRIAL: NCT01485783
Title: Improving Outcomes for Hypertensive Children
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: ABPM Hypertensive Children
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — none collected
Oversight: Data Monitoring Committee: No

SUMMARY:
Approximately 200 children age 6 - <18 years receiving medications for essential hypertension (HTN) will be recruited from the Pediatric Hypertension Clinic at the time of a routine clinic visit. Participating subjects will be asked to wear the ambulatory blood pressure monitor (ABPM) for 24 hours within 2 weeks of the qualifying visit. Measurements obtained with the ABPM will be compared to measurements obtained by routine clinical procedures documented in the subject's clinical chart. Kappa statistic will be utilized to compare differences in documented BP control between the two measures as well as changes in therapeutic management decisions by treating physicians with the addition of the ABPM readings. The overall goal is to confirm that ABPM leads to an increased detection of uncontrolled HTN along with a similar increase in adjustments increasing anti-hypertensive medication regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-17 years (up to 18th birthday) receiving anti-hypertensive medication(s) by subject history at presentation for the qualifying clinic visit
2. Arm circumference measurement of 15-50 cm (limits of SpaceLabs ABPM cuffs).

Exclusion Criteria:

1. Severe HTN which in the opinion of the treating physician would prevent the subject from delaying changes in therapy to complete the study.
2. Secondary HTN from all causes (excluding obesity-related HTN). This includes but is not limited to renovascular HTN, chronic kidney disease, coarctation of the aorta, and monogenic forms of HTN.
3. Physical limitations prohibiting placement of the ABPM monitor.
4. Significant arrhythmias or known disruptions in cardiac output which may interfere with the monitor's ability to detect BP accurately.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Approximately 200 children age 6 - <18 years receiving medications for essential HTN will be recruited from the Pediatric Hypertension Clinic at the time of a routine clinic visit.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Redwine, MD, Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States